CLINICAL TRIAL: NCT00975312
Title: Solar Lentigines Treatment With the Triple Combination Cream (Hydroquinone 4%, Tretinoin 0.05%, and Fluocinolone Acetonide 0.01%). Randomized, Double Blind, Controlled Trial.
Brief Title: Solar Lentigines Treatment With the Triple Combination Cream
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: William Andrés Romero, Pontificia Universidad Católica de Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEN-TriC-001
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Lentigo
Keywords: lentigo; hydroquinone; tretinoin; fluocinolone acetonide
MeSH Terms: conditions — Lentigo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triple combination cream (Experimental): The triple combination cream (hydroquinone 4%, tretinoin 0.05%, and fluocinolone acetonide 0.01%) was applied on the whole back of one hand.
  Interventions: Drug: Triple combination cream; Drug: Tretinoin 0.05%

INTERVENTIONS:
Drug: Triple combination cream — The triple combination cream (hydroquinone 4%, tretinoin 0.05%, and fluocinolone acetonide 0.01%) was applied on the whole back of one hand once daily for up 12 weeks.
  Other Names: Tri-luma
Drug: Tretinoin 0.05% — Tretinoin 0.05% cream was applied on the whole back of the other hand once daily for up 12 weeks.
  Other Names: Retacnyl

SUMMARY:
Background

* Lentigines are usually the first sign of photoaging and may produce a significant impact on patients' quality of life.
* There is no a treatment of choice for this condition.
* Solar lentigines and melasma share similar physiopathologic characteristics.
* The triple combination (TC) cream (hydroquinone 4%, tretinoin 0.05%, and fluocinolone acetonide 0.01%) has been effective and safe for the treatment of melasma and other hyperpigmented lesions.

Hypothesis

* The TC cream will be effective and safe for the treatment of solar lentigines on the back of the hands.

Patients and methods

* 22 patients with solar lentigines were selected and their right hand or left hand were selected at random to be treated with either TC cream or tretinoin 0.05% cream once daily for up 12 weeks.
* Patients were instructed to apply both creams on the whole back of the hand and not only in the lentigines, and to use a broad-spectrum sunscreen (SPF 50+, UVA-PF 28) daily in both hands.
* Clinical assessments of Target Lesion Pigmentation, Physician's Global Assessment of Improvement and a Subject's Self-Assessment questionnaire were collected for data analysis at weeks 4, 8, and 12 after starting the treatment and 3 month post-treatment.
* Statistical methods: The ordinally scaled efficacy measures underwent rank transformation and were analyzed by analysis of variance to test the null hypothesis of no differences among treatments. We performed Mann-Whitney and Wilcoxon tests and the XLSTAT 2009 software was used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes of 30 - 80 years of age.
* Phototype II-V.
* Postmenopausal women of childbearing age or users of any contraception method with negative pregnancy test (beta subunit chorionic gonadotropin in the blood) at baseline and that maintain the contraceptive treatment during the investigation.
* Subjects with more than 10 solar lentigines on the back of each hand wich were no treated in the last 6 months

Exclusion Criteria:

* Patients under 30 or over 80 years of age.
* Skin types I and VI.
* Less than 10 solar lentigines on the back of each hand.
* Patients who have received or are receiving any other treatment for lentigines of the back of hands.
* Women of childbearing age without contraceptive therapy.
* Pregnancy or lactation.
* History of hypersensitivity to any component of the drugs.
* Simultaneous use of other topical skin lightening.
* Patient refusal to participate in the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Target lesion pigmentation becomes equal or slightly darker than the surrounding skin | 3 months

SECONDARY OUTCOMES:
Improvement in physician's global assessment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William A Romero, MD, Principal Investigator — Pontificia Universidad Catolica de Chile; Emilia M Zegpi, MD, Study Chair — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Fleischer AB Jr, Schwartzel EH, Colby SI, Altman DJ. The combination of 2% 4-hydroxyanisole (Mequinol) and 0.01% tretinoin is effective in improving the appearance of solar lentigines and related hyperpigmented lesions in two double-blind multicenter clinical studies. J Am Acad Dermatol. 2000 Mar;42(3):459-67. doi: 10.1016/s0190-9622(00)90219-6. PMID 10688717
- [Background] Draelos ZD. The combination of 2% 4-hydroxyanisole (mequinol) and 0.01% tretinoin effectively improves the appearance of solar lentigines in ethnic groups. J Cosmet Dermatol. 2006 Sep;5(3):239-44. doi: 10.1111/j.1473-2165.2006.00260.x. PMID 17177746
- [Background] Palumbo A, d'Ischia M, Misuraca G, Prota G. Mechanism of inhibition of melanogenesis by hydroquinone. Biochim Biophys Acta. 1991 Jan 23;1073(1):85-90. doi: 10.1016/0304-4165(91)90186-k. PMID 1899343
- [Background] Petit L, Pierard GE. Analytic quantification of solar lentigines lightening by a 2% hydroquinone-cyclodextrin formulation. J Eur Acad Dermatol Venereol. 2003 Sep;17(5):546-9. doi: 10.1046/j.1468-3083.2003.00808.x. PMID 12941090
- [Background] Weinstein GD, Nigra TP, Pochi PE, Savin RC, Allan A, Benik K, Jeffes E, Lufrano L, Thorne EG. Topical tretinoin for treatment of photodamaged skin. A multicenter study. Arch Dermatol. 1991 May;127(5):659-65. PMID 2024983
- [Background] Gupta AK, Gover MD, Nouri K, Taylor S. The treatment of melasma: a review of clinical trials. J Am Acad Dermatol. 2006 Dec;55(6):1048-65. doi: 10.1016/j.jaad.2006.02.009. Epub 2006 Sep 28. PMID 17097400
- [Background] Rendon M, Berneburg M, Arellano I, Picardo M. Treatment of melasma. J Am Acad Dermatol. 2006 May;54(5 Suppl 2):S272-81. doi: 10.1016/j.jaad.2005.12.039. PMID 16631968
- [Background] Taylor SC, Torok H, Jones T, Lowe N, Rich P, Tschen E, Menter A, Baumann L, Wieder JJ, Jarratt MM, Pariser D, Martin D, Weiss J, Shavin J, Ramirez N. Efficacy and safety of a new triple-combination agent for the treatment of facial melasma. Cutis. 2003 Jul;72(1):67-72. PMID 12889718
- [Background] Ferreira Cestari T, Hassun K, Sittart A, de Lourdes Viegas M. A comparison of triple combination cream and hydroquinone 4% cream for the treatment of moderate to severe facial melasma. J Cosmet Dermatol. 2007 Mar;6(1):36-9. doi: 10.1111/j.1473-2165.2007.00288.x. PMID 17348994
- [Background] Torok H, Taylor S, Baumann L, Jones T, Wieder J, Lowe N, Jarret M, Rich P, Pariser D, Tschen E, Martin D, Menter A, Weiss J. A large 12-month extension study of an 8-week trial to evaluate the safety and efficacy of triple combination (TC) cream in melasma patients previously treated with TC cream or one of its dyads. J Drugs Dermatol. 2005 Sep-Oct;4(5):592-7. PMID 16167418
- [Result] Ortonne JP, Pandya AG, Lui H, Hexsel D. Treatment of solar lentigines. J Am Acad Dermatol. 2006 May;54(5 Suppl 2):S262-71. doi: 10.1016/j.jaad.2005.12.043. PMID 16631967